CLINICAL TRIAL: NCT01074073
Title: A Phase 1, Open-Label, 2-Period, Sequential, Drug-Drug Interaction Study To Determine The Effect Of Lithium 600 Mg BID On The Safety And Pharmacokinetics Of Lurasidone 120 Mg QD In Patients With Schizophrenia Or Schizoaffective Disorder
Brief Title: Lithium Drug-Drug Interaction Study With Lurasidone HCl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1050247
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia
Keywords: Lithium DDI with Lurasidone HCl; Male/Female, Schizophrenia Patients
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium/Lurasidone (Other): Schizophrenia Patients
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — lurasidone HCl 40 mg tablets administered orally as three tablets (120 mg) once a day (QD).
  Lithium 300 mg capsules administered orally as two capsules (600 mg) twice a day (BID).
  On dosing days, breakfast will be served 30 minutes prior to the planned dosing time. Patients must consume the breakfast within 30 minutes or less. Dosing will take place 30 minutes after the start of breakfast.

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction effect between Lithium and Lurasidone HCl.

DETAILED DESCRIPTION:
To compare the steady state pharmacokinetic profile of lurasidone 120 mg QD when administered alone vs. the steady state pharmacokinetic profile of lurasidone 120 mg QD when coadministered with steady state lithium 600 mg BID.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform.
2. Females who participate in this study:

   * are unable to have children-OR-
   * are willing to remain abstinent from Day -5 until 90 days after discharge;
3. Males must be willing to remain sexually abstinent or use an effective method of birth control (e.g. condom) from Day -5 until 90 days after discharge.
4. Able and agree to remain off of prior antipsychotic medication for the duration of the study.

Exclusion Criteria:

1. Presence or history (within the last year) of a medical or surgical condition (e.g. gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
2. Positive test results within 30 days prior to the start of the study for:
3. Participated in another clinical trial or receiving an investigational product within 30 days prior to drug administration.
4. Use of concomitant medications that prolong the QT/QTc interval within 14 days prior to Day - 5 to follow-up
5. Use of a monoamine oxidase inhibitor within 21 days prior to Day 1 to Restabilization.
6. Received depot neuroleptics unless the last injection was at least 1 treatment cycle before Day -5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bussel, MD, Principal Investigator — CCT/Parexel
Locations (1):
- CCT/Parexel, Culver City, California, United States